CLINICAL TRIAL: NCT02416687
Title: Immediate Post-partum Initiation of Etonogestrel-releasing Implant: a Randomized Controlled Trial on Breastfeeding Impact
Brief Title: Etonogestrel Implant and Postpartum Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carolina Sales Vieira, Professor, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 62798
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implanon® (Active Comparator): Postpartum women into whom the etonogestrel-releasing contraceptive implant (Implanon®, N.V. Organon, Oss, Netherlands) was inserted in the first 48 h postpartum
  Interventions: Device: Implanon®
- Control group (No Intervention): Postpartum women who used no contraceptive method in the first six weeks after delivery

INTERVENTIONS:
Device: Implanon® — Postpartum women into whom the etonogestrel-releasing contraceptive implant was inserted in the first 48 h postpartum
  Other Names: etonogestrel-releasing implant (Implanon)
  Arms: Implanon®

SUMMARY:
The etonogestrel (ENG) implant inserted immediately postpartum reduces the risk of pregnancy recurrence, especially in vulnerable populations. A limitation to recommending this practice universally is the low quality of evidence on the effect of the ENG implant on breastfeeding when inserted immediately postpartum. This study is the first assessing the impact of inserting the ENG implant immediately postpartum on the amount of milk using the gold standard method for this purpose.

DETAILED DESCRIPTION:
What is known already: The ENG implant inserted immediately postpartum reduces the risk of pregnancy recurrence, especially in vulnerable populations. A limitation to recommending this practice universally is the low quality of evidence on the effect of the ENG implant on breastfeeding when inserted immediately postpartum. This study is the first assessing the impact of inserting the ENG implant immediately postpartum on the amount of milk using the gold standard method for this purpose.

Study design, size, duration: This randomized, single-blind and controlled clinical trial evaluated 24 postpartum women and their NBs and was conducted at the Women's Health Reference Center of Ribeirão Preto, Brazil. The mother-NB pairs were evaluated for six weeks postpartum.

Participants/materials, setting, methods: Twenty-four mother-NB pairs were randomized into two groups: a) Implant group: ENG-releasing implant inserted within 48 h after delivery and b) Control group: absence of contraceptive method for six weeks after delivery. Anthropometric assessments and breastfeeding questionnaires were conducted at 4-time points of the 6-week monitoring period (at study admission and on the 14th, 29th and 43rd days after randomization). Saliva samples were collected from the mother-NB pairs prior to deuterium (D2O) dose administration. Totals of 5 g and 10 g D2O were orally administered to the postpartum women on the day of randomization (day 0) and the 29th study day, respectively. New saliva samples were collected on days 1, 2, 3, 4, 13 and 14 following intake of each D2O dose. The D2O isotope ratio was assessed in saliva samples using mass spectrometry to estimate the volume of breast milk ingested by the NB (daily average expressed as mL/day).

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18 years or older who agreed to use the ENG implant as a contraceptive method,
* Body mass index (BMI) <30 kg/m2,
* Women without contraindication to breastfeeding,
* Women whose newborns were healthy, without malformations, born at term (gestational age ≥ 37 weeks), with appropriate weight for gestational age and with normal sucking ability, were included.
* The subjects had to live in Ribeirão Preto and to have breastfed a child from a previous delivery for at least 3 months.

Exclusion Criteria:

* Tobacco smokers, drug addicts or alcoholics,
* Women with educational levels lower than 5 years,
* Women with clinical conditions considered category 3 and 4 for implant use (except insertion immediately postpartum) by the WHO (World Health Organization, 2009),
* Women with histories of psychiatric illness,
* Women using medications that could alter the concentration of etonogestrel,
* Women with known allergies to the local anesthetic lidocaine (used to place the implant),
* Women who wanted to keep their cyclic menstrual bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
breast milk intake | Six weeks after delivery
  The primary outcome was the amount of breast milk intake by the NBs through breastfeeding in the first six weeks after delivery

SECONDARY OUTCOMES:
Exclusive breastfeeding | Six weeks after delivery
  Rate of exclusive breastfeeding
Newborn weight | Six weeks after delivery
  Weight gain by newborns in six weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinica de Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil